CLINICAL TRIAL: NCT04478656
Title: Phase 1, Multicenter, Double-Blind, Placebo-Controlled, Randomized Clinical Trial to Evaluate 2 Doses of 3 Sequentially Escalating Cohort of BBV121 in Healthy Adult Dengue Sero-Negative and Dengue Sero-Positive Volunteers
Brief Title: Safety and Immunogenicity of BBV121
Acronym: Zika
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bharat Biotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BBIL/ZIKV/I/2016
Record Dates: First submitted 2017-07-17; First posted 2020-07-21 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Zika Virus Infection
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to sequential escalating dose level groups to receive vaccinations at 2.5 µg, 5 µg, or 10 µg or Placebo on Day 0 and 28 with follow-up for 12 months from initial administration of the investigational product.
Who Masked: Participant, Investigator
Masking Description: Blinded vial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BBV121-2.5 µg (Experimental): BBV121: Each 0.5ml vial contain purified10 µg inactivated Zika virus, alum, 2-PE and phosphate buffered saline qs to 0.5mL
  Interventions: Biological: BBV121
- Placebo (Placebo Comparator): Each 0.5ml vial contain purified 2.5 µg, 5 µg or 10 µg inactivated Zika virus, alum, 2-PE and phosphate buffered saline qs to 0.5mL
  Interventions: Biological: BBV121
- BBV121-5 µg (Experimental): BBV121: Each 0.5ml vial contain purified inactivated Zika virus, alum, 2-PE and phosphate buffered saline qs to 0.5mL
  Interventions: Biological: BBV121
- BBV121-10 µg (Experimental): BBV121: Each 0.5ml vial contain purified inactivated Zika virus, alum, 2-PE and phosphate buffered saline qs to 0.5ml
  Interventions: Biological: BBV121

INTERVENTIONS:
Biological: BBV121 — BBV121 or Placebo are administered intramuscularly in deltoid region on Day 0 and 28
  Other Names: Placebo

SUMMARY:
To evaluate the safety, tolerability, and immunogenicity of two-doses of three-sequentially escalating cohort (2.5 µg, 5 µg and 10 µg) of BBV121 (purified inactivated adsorbed Zika virus vaccine) compared with Placebo (Alum). The investigational product is administered intramuscularly on Day 0 and 28 with safety and immunogenicity testing on Day 0, 28 and 56, and Month 6, 9 and 12

DETAILED DESCRIPTION:
A phase 1, multicenter, double-blind, placebo-controlled, randomised (intra group) clinical trial to evaluate the safety, tolerability and immunogenicity of two-doses of three-sequentially escalating cohort (2.5 µg, 5 µg and 10 µg) of BBV121 (inactivated adsorbed Zika Virus Vaccine) compared with Placebo (Alum) administered intramuscularly on Day 0 and 28 in healthy adult Dengue Sero-Negative (Group 1) and Dengue Sero-Positive (Group 2) male and female volunteers.

Participants will be assigned to sequential escalating dose level groups to receive vaccinations at 2.5 µg, 5 µg, or 10 µg or Placebo on Day 0 and 28 with follow-up for 12 months from initial administration of the investigational product.

Immunogenicity testing on Day 0, 28 and 56, and post-study at the end of Month 6, 9 and 12 after the initial administration of the investigational product.

Safety tests (laboratory and clinical investigations) will be done during Screening, Day 0, 28, 56, and post-study at Month 6, 9 and 12 months after the initial administration of the investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy male and female volunteers aged between 18 and 65 years weighing at least 50kgs of body weight
2. Ability to comprehend the full nature and purpose of the study, including possible risks and adverse events; ability to co-operate with the Investigator and to comply with the requirements of the entire study
3. Signed written informed consent prior to inclusion in the study
4. Seronegative for Zika by ELISA
5. Dengue sero-negative at baseline by screening laboratory evaluation, confirmed by Dengue IgG by ELISA method for Group 1 participants
6. Dengue seropositive at baseline by screening laboratory evaluation, confirmed by Dengue IgG by ELISA method for Group 2 participants
7. Dengue vaccination or suffered from Dengue viral fever for Group 2 volunteers
8. No history of yellow fever vaccination
9. No history of vaccination to Japanese encephalitis vaccination
10. Since active (live) ZIKV infection is known to cause teratogenicity, women of child-bearing potential should agree to use medically effective contraception (oral contraception, barrier methods, spermicide, etc.), preferably double contraception or have a partner who is sterile from enrollment to 3 months following the last injection, or have a male partner who is medically unable to induce pregnancy.
11. Sexually active men who are considered sexually fertile must agree to use either a barrier method of contraception, preferably double contraception during the study, and agree to continue the use for at least 3 months following the last injection, or have a partner who is permanently sterile or is medically unable to become pregnant.
12. A negative urine or serum pregnancy test before administration of investigational vaccine on day of screening (Serum Pregnancy Test), and Day 0 and Day 28 (both days Urine Pregnancy Test)
13. No history of clinically significant immunosuppressive or autoimmune disease.
14. Laboratory investigations must be within normal limits

    1. Hemoglobin >10gm/dL
    2. WBC (white blood cells) >4000/mm3
    3. Platelets >100,000/mm3
    4. Bilirubin and AST/ ALT <1.5 x ULN (upper limit of normal)
    5. Creatinine <1.5 x ULN for the clinical laboratory
15. Not currently or within the previous 4 weeks taking immunosuppressive agents (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or corticosteroids at a dose less than 20 mg/day).
16. Patients should be otherwise healthy as determined by physical examination, medical history, and no significant abnormality in any of the clinical parameters including ECG and Chest X-ray.
17. Willing to allow storage and future use of biological samples for Zika virus related research.

Exclusion Criteria:

1. Administration of an investigational vaccine or drug either currently or within 30 days of first BBV121 vaccination
2. Previous receipt of an investigational vaccine or drug for the treatment or prevention of Zika virus
3. Administration of any vaccine within 4 weeks of first dose
4. Administration of any monoclonal or polyclonal antibody product within 4 weeks of the first dose of BBV121 vaccination
5. Administration of any blood product within 3 months of first dose
6. Pregnancy or breast feeding or plans to become pregnant during the study
7. Positive serologic test for HIV, hepatitis B surface antigen (HBsAg); or any potentially communicable infectious disease as determined by the Principal Investigator or Medical Monitor
8. Positive serologic test for hepatitis C (exception: successful treatment with confirmation of sustained virologic response);
9. Chronic liver disease or cirrhosis
10. Immunosuppressive illness including hematologic malignancy, history of solid organ or bone marrow transplantation
11. Current or anticipated concomitant immunosuppressive therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or corticosteroids at a dose less than 20 mg/day)
12. Current or anticipated treatment with TNF-alpha inhibitors such as infliximab, adalimumab, and etanercept
13. Prior major surgery or any radiation therapy within 4 weeks of enrolment
14. Any pre-excitation syndromes, e.g., Wolff-Parkinson-White syndrome
15. Presence of a cardiac pacemaker or automatic implantable cardioverter defibrillator
16. Metal implants within 20 cm of the planned site(s) of injection
17. Presence of keloid scar formation or hypertrophic scar at the planned site(s) of injection
18. Prisoner or participants who are compulsorily detained (involuntary incarceration) for treatment of either a physical or psychiatric illness
19. Active addictive drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements or assessment of immunologic endpoints
20. Blood donations/ losses within 2 months of screening
21. Significant orthostatic hypotension (i.e., a drop in systolic blood pressure of 30 mm Hg or more and/or a drop in diastolic blood pressure of 20 mmHg or more on standing)
22. Prior radiotherapy in 30 days or less
23. Significant pre-existing co-morbidities i. Cardiovascular

    * Myocardial infarction within the last 6 months
    * Congestive heart failure
    * Unstable angina
    * Active cardiomyopathy
    * Cardiac arrhythmia
    * Uncontrolled hypertension
    * History of familial long QT syndrome or sudden cardiac death ii. Pulmonary disease requiring oxygen iii. Neurologic and psychiatric
    * History of significant neurologic or psychiatric disorder that would preclude study compliance or ability to give informed consent iv. Rheumatic arthralgia
24. Participants not having adequate hematologic reserve i. Hemoglobin <10gm/dL ii. WBC (white blood cells) <4000/mm3 iii. ANC (absolute neutrophils count) <2000/ mm3 iv. Platelets <100,000/mm3
25. Inadequate hepatic function at screening as defined by:

    i. Bilirubin >1.5 x ULN (upper limit of normal) ii. AST/ ALT >1.5 x ULN
26. Inadequate renal function at screening as defined by:

    i. Creatinine >1.5 x ULN for the clinical laboratory
27. An unusual or abnormal diet, for whatever reason e.g. religious fasting
28. Any illness or condition that in the opinion of the investigator may affect the safety of the participant or the evaluation of any study endpoint

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-06-03 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events and Serious Adverse events | Within 2 hrs
  safety
  * Incidence of solicited AEs post-vaccination
  * Incidence of unsolicited AEs post-vaccination
  * Incidence of SAE
Occurrence of adverse events and Serious Adverse events | 7 Days
  safety
Occurrence of adverse events and Serious Adverse events | 12 months
  safety

SECONDARY OUTCOMES:
Geometric mean titre estimated by 50% plaque reduction neutralization test and four-fold seroconversion | Day 0
  Immunogenicity
Geometric mean titre estimated by 50% plaque reduction neutralization test and four-fold seroconversion | Day 28
  Immunogenicity
Geometric mean titre estimated by 50% plaque reduction neutralization test and four-fold seroconversion | Day 56
  Immunogenicity
Geometric mean titre estimated by 50% plaque reduction neutralization test | Day 365
  Immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Sudhakar Bangera, Study Chair — Bharat Biotech International Limited
Locations (1):
- Bharat Biotech International Ltd, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No